CLINICAL TRIAL: NCT05012553
Title: The Effect of Self and Peer Assesment Education Given to Nursing Students: Stoma Care
Brief Title: The Effect of Self and Peer Assesment Education Given to Nursing Students: Stoma Care Skill Example
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olga Incesu, Phd student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Florence Nightingale Faculty
Record Dates: First submitted 2021-08-02; First posted 2021-08-19 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Assessment, Self; Stoma Colostomy; Achievement
Keywords: stoma care; peer assesment; self assesment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no education about self and peer assesment (No Intervention): Stoma care skills of the group who did not receive self- and peer-assessment training will be evaluated.
- education of self and peer assesment (Experimental): Stoma care skills of the group who received self and peer assessment training will be evaluated.
  Interventions: Other: education of self and peer assesment

INTERVENTIONS:
Other: education of self and peer assesment — Stoma care skill achievement is expected to be higher in the group that received self- and peer-assessment training compared to the group that did not receive training.
  Arms: education of self and peer assesment

SUMMARY:
Self- and peer-assessment is one of the important methods among student-centered assessment methods. The ability of the student to evaluate himself and his peers provides many contributions to him in his education and professional life.Nursing education aims to gain many psychomotor skills.Aim is to examine the effects of self and peer assessment training on the success of stoma care skills.

DETAILED DESCRIPTION:
There are different results regarding the effects of self-assessment and peer assessment on psychomotor skill achievement. It is thought that the reason for this difference in results may be student-related reasons or may be related to the effectiveness of the education.

The aim is to measure the stoma care skill success of the students who are given self and peer assessment training through the rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Istanbul University-Cerrahpaşa Florence Nightingale Faculty of Nursing 1st year AGNO score not to be below 1.8
* To be registered in the HMSR 2016 Surgical Diseases Nursing course in the spring semester of the 2019-2020 academic year
* Not having received peer and self-assessment training before
* Having no previous stoma care training
* Not working as a part-time or full-time nurse

Exclusion Criteria:

* To have training in stoma care
* Having received self- and peer-assessment training
* Working as a part-time or full-time nurse
* Having an AGNO score below 1.8

Ages: 19 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
The self and peer assessment scale | Baseline,:6 months Change from self and peer assessment scale score at 6 months
  The self and peer assessment scale consists of 13 items. The scale measures the learner's tendency to self and peer assessment.A minimum score of 13 and a maximum of 65 points can be obtained from the scale. In the scale applied before and after the self and peer assessment training, the increase in the scale score of the student after the training compared to the pre-training indicates that the learner develops a positive attitude towards self and peer assessment, while the decrease in the score indicates that he develops a negative attitude. shows
self and peer assessment impressions scale | 6 months
  The scale of impressions on self and peer assessment consists of 12 items. It is applied after the self and peer assessment training.A minimum of 12 and a maximum of 60 points can be obtained from the scale. As the scale score increases, it will be thought that the learner develops a positive attitude towards self and peer assessment.
The stoma care rating scale | 6 months
  The stoma care rating scale consists of 23 items. Students who have or have not received self and peer assessment training perform stoma care through this scale and their care skills are scored with this scale.A minimum score of 0 and a maximum of 46 can be obtained from the scale. An increase in the scale score indicates that stoma care skills are improving.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Ulupınar, PhD, Study Director — Istanbul University-Cerrakpasa
Locations (1):
- Florence Nightingale Faculty of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No